CLINICAL TRIAL: NCT00917137
Title: Transbronchial Needle Aspiration in the Diagnosis of Peripheral Pulmonary Malignancy: Yield and Predictors of a Positive Aspirate
Brief Title: Transbronchial Needle Aspiration in the Diagnosis of Peripheral Pulmonary Malignancy
Status: Completed | Type: Observational
Sponsor: Maggiore Bellaria Hospital, Bologna (Other)
Responsible Party: Marco Patelli, Maggiore Bellaria Hospital
Other Study IDs: 02-Trisolini
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Pulmonary Nodule; Pulmonary Mass
Keywords: Lung cancer; Lung nodule; Transbronchial needle aspiration; Transbronchial lung biopsy; Bronchoscopy
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoalveolar Lavage Fluid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peripheral pulmonary lesions
  Interventions: Procedure: TBNA + transbronchial lung biopsy + bronchial washing

INTERVENTIONS:
Procedure: TBNA + transbronchial lung biopsy + bronchial washing

SUMMARY:
The main purposes of this study are to assess the performance characteristics of transbronchial needle aspiration (TBNA) in the diagnosis of peripheral pulmonary lesions, and to identify the predictor variables of a positive aspirate.

DETAILED DESCRIPTION:
In a recent systematic literature review (Rivera PM, Mehta AC; Chest 2007; 132: 1318-1488) TBNA showed the highest sensitivity in the diagnostic bronchoscopic approach to peripheral pulmonary lesions, as compared to the other available sampling techniques (transbronchial biopsy, brushing, washings). However, the Authors conclude that the data regarding TBNA in this setting deserve cautious interpretation because of the limited number of studies and the large differences in sample size). We designed the present study to assess the performance characteristics of TBNA, alone and in comparison with those of transbronchial biopsy, in the diagnosis of peripheral pulmonary lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Pulmonary nodule (< 3 cm) or mass (> 3 cm) at computed tomography

Exclusion Criteria:

* Refusal to sign informed consent
* Uncontrolled coagulopathy
* Pregnancy

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with pulmonary nodule or mass referred for bronchoscopy to the Thoracic Endoscopy Unit of Maggiore Hospital (Bologna Italy)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Assess sensitivity, specificity and accuracy of TBNA in the diagnosis of peripheral pulmonary lesions | 1 year

SECONDARY OUTCOMES:
Evaluate the predictor variables associated with a positive TBNA result | 1 year
Compare the performance characteristics of TBNA and transbronchial lung biopsy | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Maggiore Hospital, Bologna, Italy